CLINICAL TRIAL: NCT00097175
Title: The Effects of Mood and Tryptophan Depletion on the Neural Correlates of Affective Shifting in Mood Disorders
Brief Title: Effects of Tryptophan Depletion on Brain Processing of Emotions in Patients With Mood Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050035; 05-M-0035
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-01-15

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Serotonin; Functional MRI; Genotype; Negative Affect; MDD; Healthy Volunteer; HV
MeSH Terms: conditions — Depressive Disorder, Major

SUMMARY:
This study will investigate how the brain process emotions in healthy people and in patients who have major depression in order to better understand the causes of depression. It will examine what happens in the brain when a person responds to words related to different emotions while the brain's ability to manufacture a chemical called serotonin is reduced. Serotonin regulates functions such as emotion, anxiety and sleep, and stress hormones such as cortisol. In this study, participants' serotonin levels are reduced by depleting tryptophan, an amino acid that is the main building block for serotonin.

Healthy volunteers and patients with major depression that has been in remission for at least 3 months may be eligible for this study. Candidates must be between 18 and 50 years of age and right-handed. They are interviewed about their medical and psychiatric history, current emotional state and sleep pattern, and family history of psychiatric disorders. Screening also includes psychiatric interviews and rating scales, neuropsychological tests, physical examination, electrocardiogram (EKG), and blood, urine, and saliva tests. Women have their menstrual phase determined by a blood test and home urine ovulation test kit.

The study involves two clinic visits in which participants undergo tryptophan depletion and magnetic resonance imaging (MRI). Subjects arrive at the NIH Clinical Center in the morning after fasting overnight. They fill out questionnaires have a blood sample drawn, and then take 74 capsules that contain a mixture of amino acids found in the diet. At one visit they are given capsules that contain a balanced mixture of amino acids one would normally eat in a day; at the other visit, some of the capsules contain lactose instead of tryptophan, causing tryptophan depletion. At 2 p.m. participants fill out the same questionnaires they completed at the beginning of the day and have another blood sample drawn. Then they do a computerized test in the MRI scanner. MRI uses a magnet and radio waves to obtain pictures of the brain. For the test, subjects lie on a narrow bed that slides into the cylindrical MRI scanner. They are asked to press a button in response to words associated with different emotions that appear on a screen. Arterial spin labeling - a test that uses magnetism to measure blood flow in different areas of the brain-is also done during the procedure. After the scan, subjects eat a meal and then return home.

DNA from the participants' blood samples is also examined to try to better understand the genetic causes of depression. Some of the white cells from the samples may also be grown in the laboratory so that additional studies can be done later.

...

DETAILED DESCRIPTION:
Major depressive disorder (MDD) has been associated with abnormally reduced function of central serotonergic systems by various types of evidence. One instructive paradigm for investigating the relationship between serotonergic function, cognition and depression has involved the mood response to tryptophan depletion (TD), achieved by oral loading with all essential amino acids excepting the 5-HT precursor, tryptophan. Subjects who are depressed show altered behavioral and neural response to affectively valenced stimuli, similar to those seen under TD.

More, specifically, increased response latencies to happy words have been noted in both depressed patients and healthy controls following TD using the Affective Go/No go (AGNG) test, in which subjects are required either to respond or inhibit a response to a series of emotionally valenced words.

The first round of our study employed fMRI imaging of BOLD response and arterial spin labeling to investigate response to affectively valenced words under TD in two groups, remitted MDD (rMDD) patients and healthy controls with no family history of depression. We have thus far examined the effects of TD depletion in our healthy control group. We found that emotional information processing was indeed altered by 5-HT depletion.

A behavioral bias toward positive stimuli was attenuated following depletion, which was accompanied by increased hemodynamic responses during the processing of emotional words in several subcortical structures, including the ventral striatum, hippocampal cortex, anterior insula, superior temporal gyrus and posterior cingulate. Further, inter-individual differences in tryptophan depletion-elicited anxiety correlated positively with caudate bias toward negative stimuli. On the basis of these data, we suggest that the bias towards positive stimuli might represent a normal suppression of attention to negative stimuli; a process which is abrogated in conditions, such as depression, which are characterized by a serotonergic dysfunction. In the second round of this study, we are examining whether such biases also occur beneath the level of conscious awareness.

One of the weaknesses of these data is that the patients were consciously aware of the verbal stimuli that were presented to them and likely possess learned, individualized associations to the verbal stimuli in question. We have developed a conditioning task which obviates this problem through the presentation of emotionally-valenced visual stimuli below the threshold of conscious awareness.

Since embarking on the first two phases of this study, a new paradigm has been developed which may provide further insight into affective behavioral biases. The Split Reversals task is a pavlovian reversal-learning task which allows the assessment of responses to expected and unexpected punishment and reward cues. Previous research with this task has demonstrated that reduction of serotonin in healthy individuals removes a disproportionate inability to predict punishment at baseline. In other words, serotonin reduction removes a positive bias on this task. . This is consistent with the observed removal of a positive bias on the AGNG following TD. However, on the split reversals task this positive bias is revealed by an inability to process negative stimuli at baseline, which is improved, rather than a bias towards positive stimuli which is diminished, by TD. As such, the new task provides a different direction from which to consider the emotional biases observed in affective disorders. We have suggested that the bias on the new task reflects a serotonin-mediated suppression of responses to negative stimuli in healthy individuals which, in turn, promote resilience to affective disorders. Serotonin reduction via TD hence removes this bias. That this task may therefore be sensitive to cognitive biases resulting from resilience mechanisms.

Similarly, fear potentiated startle which has been shown to be sensitive to the symptoms of anxiety has been shown to be reduced by the elevation of 5-HT via two week citalopram treatment. This is consistent with reduced processing of negative information following 5-HT increase (Grillon et al 2009). We predict that reducing 5-HT via TD will have the opposite effect and increase the duration of fear potentiated startle processing. This would provide an indirect link between reduced 5-HT and anxiety disorders. As such, we include this task in a new phase of this protocol.

In addition these behavioural TD findings, this task has been neuroimaged (fMRI) in healthy individuals. As predicted, the striatum was shown to be involved in reward processing, whilst the amygdala was shown to be involved in punishment processing. A subproject of this study will therefore attempt to extend the prior findings from the split reversals task (and reconcile them with the AGNG findings) by examining healthy individuals completing the task whilst undergoing both serotonin manipulation (TD) and fMRI. This subproject will be initially restricted to healthy individuals and should provide us with further insight into the neural substrates involved in serotonergic inhibition of aversive processing highlighted by the first phase of this study. This will also provide a basis from which to consider potential future study with the same task in MDD subjects undergoing TD.

There may well be a genetic basis to these phenomena. It is known that the functional variant in the promoter region of the serotonin transporter gene (5-HTTLPR) is partly responsible for determining how individuals respond to TD. In fact, recently reported that carriers of the short 5-HTTLPR allele showed impaired recognition of fearful faces following TD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers

Right-handed subjects (ages 18-50) will be selected who have not met criteria for any major psychiatric disorder, have no known first-degree relatives with mood disorders, and have a current score on the Hamilton Depression Rating Scale (HDRS; 17 item) in the not depressed range ( 7). Control subjects will be matched to depressed subjects and their relatives for age, gender, and education.

MDD Samples

Right-handed subjects (ages 18-50) will be selected with a past history of MDD by DSM-IV criteria.

Healthy Relatives

Healthy, right-handed, first-degree relatives of patients with MDD will be recruited.

EXCLUSION CRITERIA:

Subjects must not have taken antidepressant drugs for at least 3 months (4 months for fluoxetine) prior to the fMRI studies or other medications likely to alter monoamine neurochemistry or cerebrovascular and cardiovascular function for at least 3 weeks prior to imaging. However, effective medications will not be discontinued for the purposes of this study. Subjects will also be excluded if they have:

1. Psychosis
2. Medical or neurological illnesses likely to affect physiology or anatomy, i.e. hypertension, cardiovascular disorders
3. A history of drug (including benzodiazepines (BZD)) abuse within 1 year or a lifetime history of drug dependence (DSM IV criteria)
4. A history of alcohol abuse within 1 year or a lifetime history of alcohol dependence (DSM IV criteria)
5. Current pregnancy (as documented by pregnancy testing at screening or at days of the challenge studies)
6. Current breast feeding
7. Are smokers
8. Serious suicidal ideation or behavior. In this study, there is a small risk of transient depressive symptoms occurring after ingesting the amino acid mixture. Therefore, if volunteers manifest evidence of serious suicidal ideation or behavior, they will be excluded from participating. Criteria for meeting suicidal ideation include but are not limited to: 1) thoughts of suicide within the past 3 months which are accompanied by intent to harm oneself, serious consideration of means or plan to attempt suicide, evidence of arranging for a suicide attempt (e.g. giving away prized possessions or updating a will), or clear desire to commit suicide, 2) severity of past suicide events, if applicable or 3) a current plan for harming themselves. All assessments will be conducted by an experienced, NIMH credentialed health professional, such as a psychiatrist or psychiatric nurse who will use their expert knowledge and experiences in determining the authenticity of a participant s information and handle the situation accordingly.
9. General MRI exclusion criteria

Subjects must exhibit no or only moderate alcohol use. Subjects with current or previous regular use (greater than 4 weeks) of BZDs and excessive use of alcohol (greater than 8 ounces/day for men and greater than 6 ounces/day for women) in the past or present are ineligible for participation, as such drug use may confound the results. Smokers (regular use within the last 3 months) are ineligible because of the evidence for interactions between nicotine and depression, and the possibility of withdrawal symptoms that may affect behavioral and neural responses to TD.

Subjects beyond age 50 are excluded to address the biological heterogeneity encompassed by the MDD criteria, since depressives whose age-at-onset is later than 50 have a far greater likelihood of having MRI correlates of cerebrovascular disease than age-matched healthy controls or age-matched early-onset depressives. Subjects whose first major depressive episodes arose temporally after other medical or psychiatric conditions will also be excluded, since their functional imaging results generally differ from those reported in primary MDD.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2004-11-10; Study Completion 2014-01-15

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grillon, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Drevets WC, Price JL, Simpson JR Jr, Todd RD, Reich T, Vannier M, Raichle ME. Subgenual prefrontal cortex abnormalities in mood disorders. Nature. 1997 Apr 24;386(6627):824-7. doi: 10.1038/386824a0. PMID 9126739
- [Background] Lesch KP, Bengel D, Heils A, Sabol SZ, Greenberg BD, Petri S, Benjamin J, Muller CR, Hamer DH, Murphy DL. Association of anxiety-related traits with a polymorphism in the serotonin transporter gene regulatory region. Science. 1996 Nov 29;274(5292):1527-31. doi: 10.1126/science.274.5292.1527. PMID 8929413
- [Background] Moreno FA, Rowe DC, Kaiser B, Chase D, Michaels T, Gelernter J, Delgado PL. Association between a serotonin transporter promoter region polymorphism and mood response during tryptophan depletion. Mol Psychiatry. 2002;7(2):213-6. doi: 10.1038/sj.mp.4000962. PMID 11840315